CLINICAL TRIAL: NCT06758908
Title: Prevelance, Predictors and Outcome of Sepsis Associated Liver Injury (SALI)
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Collaborators: Investigator (Unknown)
Responsible Party: Principal Investigator, Mahmoud sayed Zohry Sayed, assiut university, Assiut University
Other Study IDs: prevelance ,predictors of SALI
Record Dates: First submitted 2024-12-14; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Liver Injuries
MeSH Terms: interventions — Antibiotic Prophylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SALI
  Interventions: Device: Antibiotic

INTERVENTIONS:
Device: Antibiotic — SALI

SUMMARY:
prevelance, predictors and outcome of sepsis associated liver injury (SALI)

DETAILED DESCRIPTION:
patient with liver disease and sepsis at the same time

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of SALI
* must take liver support

Exclusion Criteria:

* SALI
* Thyroid disease

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all people between 15 to 75 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
prevelance, predictors and outcome of sepsis associated liver injury (SALI) | baseline
  analysis outcome of sepsis associated liver injury (SALI)
28 days mortality | baseline
  patient with liver dieases and sepsis
patient shouldn't be in pain | baseline
  patient in study not in pain

SECONDARY OUTCOMES:
patient stay in hospital 2weeks | baseline
  patient with liver dieases and sepsis

IPD SHARING:
Plan to Share IPD: No